CLINICAL TRIAL: NCT05060419
Title: Phase Ⅱ, Randomized, Double-Blind,Double-Dummy Study Evaluating Safety,Tolerability,Efficacy of Meropenem-FL058 in Adult Patients With Complicated Urinary Tract Infections, Including Acute Pyelonephritis
Brief Title: Meropenem-FL058 Phase 2 Study in the Treatment of Complicated Urinary Tract Infections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FL058-II-01
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: interventions — Piperacillin, Tazobactam Drug Combination; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind,Double-Dummy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meropenem-FL058 (180min infusion) (Experimental)
  Interventions: Drug: Meropenem- FL058; Drug: Saline
- Piperacillin-Tazobactan (30min infusion) (Active Comparator)
  Interventions: Drug: Piperacillin -tazobactam; Drug: Saline

INTERVENTIONS:
Drug: Meropenem- FL058 — Meropenem-FL058(Meropenem 1000mg plus FL058 1000mg)q8h
  Meropenem-FL058(Meropenem 2000mg plus FL058 1000mg)q8h
  Arms: Meropenem-FL058 (180min infusion)
Drug: Piperacillin -tazobactam — Piperacillin-tazobactam (piperacillin 4 g plus tazobactam 0.5 g)q8h
  Arms: Piperacillin-Tazobactan (30min infusion)
Drug: Saline — 180min
  Arms: Piperacillin-Tazobactan (30min infusion)
Drug: Saline — 30min
  Arms: Meropenem-FL058 (180min infusion)

SUMMARY:
Phase 2, randomised, double-blind,double-dummy study in hospitalised adults with complicated urinary tract infection (cUTI), including acute pyelonephritis.Treatment duration for each cohort was 7 to 14 days. Patients were not permitted to switch to oral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 18 ~ 75 years (inclusive);；
2. Acute pyelonephritis or other complicated urinary tract infection.

Exclusion Criteria:

1. Patients needing concomitant systemic antimicrobial agents in addition to those designated in the various study treatment groups;
2. Fungal urinary tract infection;
3. History of allergic to any carbapenem, cephalosporin, penicillin, other β -lactam drugs or other β -lactamase inhibitors;
4. Pregnant or breastfeeding women;
5. Inability to tolerate intravenous fluids, due to medical reasons, of 1050 mL per day required for study drug administration;
6. Unable or unwilling, in the judgment of the Investigator, to comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-08 (Estimated); Primary Completion 2022-04-29 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in the Microbiological Modified Intent to Treat (m-MITT) Population who achieve overall treatment success at Test Of Cure (TOC). | 5 to 9 days post-End of Treatment
  Treatment success is defined as the composite of clinical outcome of Cure and the microbiological outcome of Eradication.

CONTACTS AND LOCATIONS:
Overall Officials: Huang Haihui, Professor, Principal Investigator — Huashan Hospital